CLINICAL TRIAL: NCT02195778
Title: Assessment of Health Literacy Among Adult Patients in the United Arab Emirates to Facilitate Clinical Trials Recruitment.
Acronym: LIT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tawam Hospital (Other)
Responsible Party: Principal Investigator, Dr Satish Chandra, Senior Specialist, Tawam Hospital
Other Study IDs: CRD 262/13
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Health Literacy; Adult; UAE; Disease; Age
Keywords: Health Literacy; Adult; UAE; Disease; Age
MeSH Terms: conditions — Disease

STUDY DESIGN:
Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Young, 18 to 30
- Middle, 31 to 50
- Older, 51 to 70

SUMMARY:
Health Literacy is the ability to understand health information and to use that information to make good decisions about health and medical care. Health informatin can overwhelm even people with advanced literacy skills. About one third of the adult population in the United States has limited health literacy.

DETAILED DESCRIPTION:
Health literacy is the ability to understand health information and to use that information to make good decisions about health and medical care. Health information can overwhelm even people with advanced literacy skills.

About one third of the adult population in the United States has limited health literacy (Berkman ND, Davis TC, McCormack L. Health literacy:what is it? J Health Commun. 2010; 15 Suppl 2: 9-19). Initial assessment of regulatory compliance in research studies in the UAE indicated poor understanding of medical information by patients/subjects (AAMDHREC 12/55).

Health Literacy Survey (HLS) will be conducted on adults visiting the participating UAE hospitals/clinics. The survey will be conducted by a trained bilingual healthcare professional such as a team of medical residents.

The investigators study attempts to identify the population that are unable to understand health information or are impaired in their understanding of health information.

ELIGIBILITY:
Inclusion Criteria:

* 18 and above
* Willing to consent

Exclusion Criteria:

* Less than 18
* Severly ill
* Unable to consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult 18+
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Patient unable to read and write. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Tawam Hospital, Al Ain City, Abu Dhabi Emirate, United Arab Emirates